CLINICAL TRIAL: NCT04191239
Title: Two Different Types of Ventilation in Preterm Neonates; Bilevel Volume Guarantee and Pressure Regulated Volume Control
Brief Title: Comparing Two Different Modes of Ventilation in Pretem Neonates Bilevel VG and PRVC
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: 2019512-2
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2020-01

CONDITIONS: Newborn Morbidity; Respiratory Failure; Bronchopulmonary Dysplasia; Mechanical Ventilation Complication
MeSH Terms: conditions — Respiratory Insufficiency; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRVC: Preterm infants with need of mechanical ventilation will receive PRVC mode until extubation
  Interventions: Device: GE ventilator with two different modes
- Bilevel VG: Preterm infants with need of mechanical ventilation will receive Bilevel VG mode until extubation
  Interventions: Device: GE ventilator with two different modes

INTERVENTIONS:
Device: GE ventilator with two different modes — GE ventilator with two different modes

SUMMARY:
Intubated preterm infants between 800-1200 grams and under 32 weeks of gestational age will start with PRVC ventilation mode, basal blood gases and work of breathing will measured. After that mode will shift to Bilevel Volume Guarantee mode for two hours than clinical and other parameters will be checked again. After this intervention, patients will allocated to PRVC or Bilevel VG group for remaining time.

ELIGIBILITY:
Inclusion Criteria:

* Need for mechanical ventilation
* 800-1200 grams of birthweight
* Surfactant received
* under 32 weeks of gestational age

Exclusion Criteria:

No need to intubation Congenital anomalies

-

Ages: 1 Day to 3 Months | Sex: All
Age Groups: Child
Study Population: All preterms under 32 weeks and between 800-1200 grams, intubated and ventilated in neonatal intensvie care unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Intubation time | 8 weeks
  Duration of mechanical ventilation

SECONDARY OUTCOMES:
Oxygen dependency | 8 weeks
  Need for supplemantal oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No